CLINICAL TRIAL: NCT03864913
Title: Investigating the Efficacy of Subcutaneous Testosterone Compared to Intramuscular Testosterone in Gender Affirming Care of Transgender Male Adolescents
Brief Title: Comparing Subcutaneous Testosterone to Intramuscular Testosterone in Gender Affirming Care of Transgender Male Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kara Connelly, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017454
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Health Services for Transgender Persons; Transgender Persons
Keywords: Gender affirming care
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Randomized arm (SQ, IM), as well as non-randomized SQ and non-randomized IM.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized SQ vs IM (Experimental): Subjects randomized to either SQ or IM testosterone injections follow study protocol.
  Interventions: Drug: Testosterone injection; Behavioral: PedsQL questionnarie; Other: Masculinizing effects questionnaire; Other: Medication experience questionnaire
- Non-randomized SQ (Experimental): Subjects choose to participate in study, but decline to randomize and select SQ injections. Follow same study protocol.
  Interventions: Drug: Testosterone injection; Behavioral: PedsQL questionnarie; Other: Masculinizing effects questionnaire; Other: Medication experience questionnaire
- Non-randomized IM (Experimental): Subjects choose to participate in study, but decline to randomize and select IM injections. Follow same study protocol.
  Interventions: Drug: Testosterone injection; Behavioral: PedsQL questionnarie; Other: Masculinizing effects questionnaire; Other: Medication experience questionnaire

INTERVENTIONS:
Drug: Testosterone injection — SQ or IM testosterone injections for pubertal induction of transgender male adolescents. Increasing doses per protocol at 3 month and 6 month follow up.
Behavioral: PedsQL questionnarie — Validated Pediatric Quality of Life questionnaire completed by subjects at baseline, 3 month and 6 month study visits.
Other: Masculinizing effects questionnaire — Subjects complete self-reported questionnaire at 3 month and 6 month study visits.
Other: Medication experience questionnaire — Subjects complete self-reported questionnaire at 3 month and 6 month study visits.

SUMMARY:
The trial studies the efficacy of subcutaneous (SQ) testosterone compared to intramuscular (IM) testosterone therapy during the first 6 months of pubertal induction in transgender male adolescents. Describes rate of adverse effects, masculinizing effects and quality of life while receiving testosterone. Evaluates clinic utilization required for testosterone therapy.

DETAILED DESCRIPTION:
Objectives:

1. Determine the efficacy of SQ testosterone compared to IM testosterone therapy. Hypothesis: SQ testosterone is equally efficacious to IM testosterone in achieving mid-pubertal testosterone levels and masculinizing physical changes in transgender male adolescents after 6 months.
2. Determine the rate of adverse reactions of SQ and IM testosterone during the first 6 months of treatment.

   Hypothesis: SQ testosterone results in equal or fewer adverse reactions than IM testosterone.
3. Evaluate quality of life (QOL) and satisfaction of injection technique for SQ and IM testosterone.

   Hypothesis: Subjects receiving SQ testosterone will report equal or superior quality of life and satisfaction with injection technique compared to IM testosterone as SQ is less painful and easier to administer at home.
4. Evaluate and compare the number of clinical visits required for testosterone injections by transgender male patients receiving SQ and IM therapy.

Hypothesis: Subjects using SQ testosterone will have fewer clinic visits than those using IM testosterone. This may impact healthcare-related costs.

Study Outline:

6 month study consisting of three study visits at baseline, 3 months and 6 months. Optional cross over of injection modality from 6-9 months. At each visit subjects complete blood work and questionnaires to determine testosterone peak and trough levels as well as biochemical adverse effects, quality of life, masculinizing effects and medication experience.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone naive
* Transgender male
* 14-19 years old

Exclusion Criteria:

* Transgender males who have received testosterone therapy in the past

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transgender male
Enrollment: 26 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Serum testosterone level | Two lab draws, before and after testosterone injection, drawn at 3 month and 6 month follow up
  Trough and peak serum testosterone level

SECONDARY OUTCOMES:
Rate of adverse effects | Assessed at 3 month and 6 month follow up
PedsQL questionnaire score | Completed at baseline, 3 month and 6 month follow up
  Validated pediatric quality of life tool
Masculinizing effects | Completed at 3 month and 6 month follow up
  Self reported, questionnaire
Medication experience | Completed at 3 month and 6 month follow up
  Self reported, questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kara Connelly, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No